CLINICAL TRIAL: NCT05830539
Title: A Phase Ib/II, Open-label, Multicenter Clinical Study to Evaluate the Antitumor Activities, Safety, and Tolerability of IN10018 Combination Therapy in Previously-treated Locally Advanced or Metastatic Solid Tumor Patients
Brief Title: IN10018 Combination Therapy in Previously-treated Locally Advanced or Metastatic Solid Tumor Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InxMed (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN10018-010
Record Dates: First submitted 2023-03-31; First posted 2023-04-26 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Triple Negative Breast Cancer(TNBC) (Experimental): Group 1: IN10018 in combination with PLD in Subjects with previously-treated locally advanced or metastatic TNBC.
  Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with previously-treated locally advanced or metastatic TNBC.
  Interventions: Drug: IN10018+PLD; Drug: IN10018+PLD+Toripalimab
- Head and Neck Squamous Cell Cancer(R/M-HNSCC) (Experimental): Group 1: IN10018 in combination with PLD in Subjects with previously-treated R/M-HNSCC.
  Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with previously-treated R/M-HNSCC.
  Interventions: Drug: IN10018+PLD; Drug: IN10018+PLD+Toripalimab
- Platinum-resistant Ovarian Cancer (Experimental): Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with platinum-resistant ovarian cancer.
  Interventions: Drug: IN10018+PLD+Toripalimab
- Platinum-sensitive Ovarian Cancer(PSOC) (Experimental): Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with Platinum-sensitive recurrent ovarian cancer.
  Interventions: Drug: IN10018+PLD+Toripalimab
- Small Cell Lung Cancer(SCLC) (Experimental): Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with previously-treated locally advanced or metastatic SCLC.
  Interventions: Drug: IN10018+PLD+Toripalimab
- Other solid tumor (Experimental): Group 1: IN10018 in combination with PLD in Subjects with other previously-treated locally advanced or metastatic solid tumors.
  Group 2: IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in Subjects with other previously-treated locally advanced or metastatic solid tumors.
  Interventions: Drug: IN10018+PLD; Drug: IN10018+PLD+Toripalimab

INTERVENTIONS:
Drug: IN10018+PLD — IN10018 orally once daily; PLD 40mg/m2, Q4W
  Other Names: IN10018 and Doxorubicin Hydrochloride Liposome Injection
  Arms: Head and Neck Squamous Cell Cancer(R/M-HNSCC); Other solid tumor; Triple Negative Breast Cancer(TNBC)
Drug: IN10018+PLD+Toripalimab — IN10018 orally once daily; PLD 40mg/m2, Q4W; Toripalimab 3 mg/kg, Q2W
  Other Names: IN10018 and Doxorubicin Hydrochloride Liposome Injection and Toripalimab

SUMMARY:
This is a multicenter, open-label, Phase Ib/II clinical trial to evaluate the safety, tolerability, and antitumor efficacy of IN10018 in combination with pegylated liposomal doxorubicin (PLD) or IN10018 in combination with PLD and anti-PD-1 in subjects with locally advanced or metastatic solid tumors who have failed or not tolerated to at least first-line system therapy.

DETAILED DESCRIPTION:
This study is a phase Ib/II, multicenter, open-label clinical study. This study consists of 2 parts: 1) Efficacy exploration part: including phase-Ib study (dose confirmation part) and phase II study, the purpose of phase Ib-dose confirmation part is to determine the Phase II recommended dose (RP2D) of IN10018 in combination with Pegylated liposomal doxorubicin (PLD) and programmed death-1 (PD-1) monoclonal antibody. The Phase II study will explore the antitumor efficacy and safety of IN10018 in combination with PLD or IN10018 in combination with PLD and anti-PD-1 monoclonal antibody in subjects with locally advanced or metastatic solid tumors who have failed or are intolerant to at least first-line system therapy; 2) Efficacy confirmation part: The antitumor efficacy and safety of combination therapy in the corresponding solid tumors will be further confirmed.

ELIGIBILITY:
Inclusion Criteria

1. Male or female, and aged 18 - 75 years at the time of signing the informed consent.
2. Has ability to understand and willingness to sign informed consent(s).
3. Histologically confirmed locally advanced or metastatic solid tumors:

   1. Cohort 1: Histologically-confirmed Locally advanced or metastatic triple-negative breast cancer.
   2. Cohort 2: Histologically or cytologically confirmed recurrent or metastatic head and neck squamous cell carcinoma.
   3. Cohort 3 and 4: Histologically confirmed epithelia ovarian cancer, fallopian tube cancer or primary peritoneum cancer with the subtype limited to high-grade serous carcinoma (HGSC) only.
   4. Cohort 5: Histologically confirmed extensive-stage small cell lung cancer (according to the Veteran's Administration Lung Cancer Study Group (VALG) classification system).
   5. Cohort 6: other Histologically confirmed locally advanced or metastatic solid tumors except cohort 1-5.
4. Have received at least 1 line of standard therapy for locally advanced or metastatic solid tumors and have failed or are not tolerable.
5. At least one measurable lesion can be accurately measured per RECIST 1.1 as assessed by investigator.
6. ECOG performance status of 0 or 1.
7. Life expectancy of at least 3 months as assessed by investigator.
8. Adequate bone marrow, liver, renal, and coagulation function within 7 days prior to first dose of study treatment.
9. Must have recovered from all AEs due to previous therapies to ≤ Grade 1 (CTCAE 5.0) or stable status as assessed by investigator.

Exclusion criteria

1. Has had major surgery or significant traumatic injury within 28 days prior to first dose of study treatment, or diagnostic biopsies within 14 days prior to first dose of study treatment.
2. Has received prior systemic anticancer therapy such as chemotherapy, biological therapy, endocrine therapy, immunotherapy, etc. within 4 weeks before the first dose.
3. History of autoimmune disease requiring systemic therapy within the past 2 years, including but not limited to autoimmune thyroid disease, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease.
4. Has interstitial pneumonia currently.
5. Has received prior treatment of any FAK inhibitor.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
7. Has a prior history of malignancy other than the study disease.
8. Clinically symptomatic pleural effusion, pericardial effusion, or ascites, or those who have received or necessary for drainages within 3 months prior to the first dose of study treatment.
9. Has malabsorption syndrome or inability to take oral medication.
10. Has clinical or radiologic evidence of bowel obstruction, or prior recurrent bowel obstruction with the cause not eliminated within 3 months prior to the first dose of study treatment.
11. Has any active infection requiring systemic therapy within 14 days prior to the first dose of study treatment.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Known allergy or hypersensitivity to IN10018, PLD, or Toripalimab or their ingredients.
14. Pregnant or lactating women.
15. Has received prior cumulative doxorubicin or equivalent anthracyclines doses of 360 mg/m2 or more.
16. Has received systemic treatment of CYP3A4, CYP2D6 or P-gp strong inhibitors/inducers within 14 days prior to the first dose of study treatment, or anticipation of the systemic treatment of these drugs during Treatment Phase.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of IN10018 in combination with PLD and anti-PD-1 monoclonal antibody. | Up to 6 Months
  Evaluate the number of patients with dose-limited toxicities (DLTs); Determine the RP2D of IN10018 in combination with PLD and Toripalimab.
Objective response rate (ORR) per RECIST v1.1 in IN10018 combined with PLD group or in IN10018 combined with PLD and anti-PD-1 monoclonal antibody group. | Up to 24 Months
  Defined as the proportion of subjects with complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Number of patients with adverse event; Number of patients with laboratory abnormalities, abnormal vital signs and abnormal 12-lead ECG. | Up to 24 Months
  Number of patients with adverse event; Number of patients with laboratory abnormalities, abnormal vital signs and abnormal 12-lead ECG.
Duration of objective response (DOR) per RECIST v1.1 in IN10018 combined with PLD group or in IN10018 combined with PLD and anti-PD-1 monoclonal antibody group. | Up to 24 Months
  Defined as the time from start of the first documentation of CR or PR to the first documentation of disease progression or to death due to any cause, whichever comes first.
Disease Control Rate (DCR) per RECIST v1.1 in IN10018 combined with PLD group or in IN10018 combined with PLD and anti-PD-1 monoclonal antibody group. | Up to 24 Months
  Defined as the proportion of patients with CR, PR, or stable disease (SD).
Progression-free survival (PFS) per RECIST v1.1 in IN10018 combined with PLD group or in IN10018 combined with PLD and anti-PD-1 monoclonal antibody group. | Up to 24 Months
  Defined as the time from start of study treatment to first documentation of disease progression or to death due to any cause, whichever comes first.
Overall survival (OS) in IN10018 combined with PLD group or in IN10018 combined with PLD and anti-PD-1 monoclonal antibody group. | Up to 36 Months
  Defined as the time from the start of study treatment to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying WU, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Xichun Hu, Principal Investigator — Fudan University; Dongmei Ji, Principal Investigator — Fudan University
Locations (7):
- China (7):
  - Anyang Tumor Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Third Hospital of Nanchang, Nanchang, Jiangxi
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality